CLINICAL TRIAL: NCT02273752
Title: Phase II Evaluation of Real-Time, Pharmacokinetically Guided Everolimus in Patients With Hormone Receptor Positive Breast Cancer, Pancreatic Neuroendocrine Tumors (PNET), and Renal Cell Carcinoma
Brief Title: Pharmacokinetically Guided Everolimus in Patients With Breast Cancer, Pancreatic Neuroendocrine Tumors, or Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, R. Donald Harvey, PharmD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00072091; NCI-2014-02112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP2645-14 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Gastrinoma; Glucagonoma; HER2-negative Breast Cancer; Insulinoma; Mucositis; Oral Complications; Pancreatic Polypeptide Tumor; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Recurrent Islet Cell Carcinoma; Recurrent Renal Cell Cancer; Somatostatinoma; Stage III Renal Cell Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Mucositis; Breast Neoplasms; Carcinoma, Islet Cell; Carcinoma, Renal Cell; Somatostatinoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (real-time pharmacokinetic TDM of everolimus) (Experimental): Patients receive everolimus PO daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo real-time pharmacokinetic TDM on days 4, 8, and 15 of course 1. Dosing adjustments of everolimus will be performed on day 8, if necessary. If the everolimus dose is adjusted, patients will continue to undergo real-time pharmacokinetic TDM weekly until goal concentrations are achieved on 2 consecutive measures. Patients whose everolimus dose is not adjusted undergo real-time pharmacokinetic TDM on day 1 of courses 2-6.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001

SUMMARY:
This phase II trial studies how well real-time pharmacokinetic therapeutic drug monitoring works in preventing stomatitis from developing in patients with hormone receptor positive breast cancer, pancreatic neuroendocrine tumors, or kidney cancer that are receiving a type of cancer drug called everolimus. Stomatitis is a common side effect of everolimus that causes inflammation of the mouth, with or without oral ulcers, and frequently leads to patients discontinuing the medication. Monitoring the blood levels of everolimus and making adjustments in a patient's dose may be able to decrease the incidence of stomatitis, while maintaining the effectiveness of everolimus to treat the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine frequency of any grade of stomatitis at day 29 (cycle 2, day 1) in patients receiving dose-adjusted everolimus.

SECONDARY OBJECTIVES:

1. Progression-free survival rates at 6 months.
2. Pharmacodynamic (PD)-inhibition of downstream mammalian target of rapamycin (mTOR) effectors in peripheral blood.
3. Number of dose adjustments required.
4. Percentage of days on therapy.
5. Average minimum concentration (Cmin) values.
6. Frequency and type of treatments for stomatitis.
7. Genetic predictors of stomatitis development in selected outlier patients.

OUTLINE:

Patients receive everolimus orally (PO) daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo real-time pharmacokinetic therapeutic drug monitoring (TDM) on days 4, 8, and 15 of course 1. Dosing adjustments of everolimus will be performed on day 8, if necessary. If the everolimus dose is adjusted, patients will continue to undergo real-time pharmacokinetic TDM weekly until goal concentrations are achieved on 2 consecutive measures. Patients whose everolimus dose is not adjusted undergo real-time pharmacokinetic TDM on day 1 of courses 2-6.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Confirmed diagnosis of:

  * Postmenopausal advanced hormone receptor-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancer after failure of treatment with letrozole or anastrozole
  * Progressive neuroendocrine tumors of pancreatic origin (PNET) that is unresectable, locally advanced or metastatic
  * Advanced renal cell carcinoma (RCC) after failure of treatment with sunitinib or sorafenib
* Histologically confirmed, measurable or evaluable disease. Patients should have at least one measurable lesion.
* Adequate bone marrow function as indicated by the following:

  * Absolute neutrophil count (ANC) > 1,500/μL
  * Platelets ≥ 100,000/μL
  * Hemoglobin > 10 g/dL
* Adequate renal function, as indicated by creatinine clearance > 30 mL/min
* Adequate liver function, as indicated by:

  * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * International normalized ratio (INR) ≤ 2
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2 x ULN unless related to primary disease
* Signed informed consent
* Adequate birth control when appropriate
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc., but not including somatostatin analogues, e.g., octreotide)
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Patients who have any severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Symptomatic congestive heart failure of New York Heart Association Class III or IV
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-DNA and/or positive HbsAg, quantifiable hepatitis C virus [HCV]-RNA)
  * Known severely impaired lung function (spirometry and diffusing capacity of the lung for carbon monoxide [DLCO] 50% or less of normal and O2 saturation 88% or less at rest on room air)
  * Active, bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed.
* Known history of HIV seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines.
* Patients who have a history of another primary malignancy, with the exceptions of: nonmelanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥3 years
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
  * Total abstinence
  * Male/female sterilization
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Donald Harvey, PharmD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited at Winship Cancer Institute of Emory University from November 2014 to December 2015.
Groups:
- Supportive Care (Real-time Pharmacokinetic TDM of Everolimus): Patients receive everolimus PO daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo real-time pharmacokinetic therapeutic drug monitoring (TDM) on days 4, 8, and 15 of course 1. Dosing adjustments of everolimus will be performed on day 8, if necessary. If the everolimus dose is adjusted, patients will continue to undergo real-time pharmacokinetic TDM weekly until goal concentrations are achieved on 2 consecutive measures. Patients whose everolimus dose is not adjusted undergo real-time pharmacokinetic TDM on day 1 of courses 2-6.
  Everolimus: Given PO
Period: Overall Study
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Trial was terminated early | 2

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Stomatitis
Description: Stomatitis graded rates and severity will be evaluated and recorded per World Health Organization and Common Terminology Criteria for Adverse Events criteria in the study population.
Time Frame: Day 29
Population: Trial was closed early due to lack of timely accrual. Because study was not fully enrolled, outcomes were unable to be measured accurately.
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be evaluated based on rates of cancer progression and time to progression in the population. Progression will be determined using standard RECIST criteria. The median PFS for this study will be estimated by Kaplan-Meier method along with 95% confidence interval.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

3. Secondary Outcome: Downstream Markers of Mammalian Target of Rapamycin (mTOR) Function Measured in Peripheral Blood Mononuclear Cells
Description: Pharmacodynamics will be evaluated for phosphorylated and non-phosphorylated ribosomal protein S6 kinase, protein kinase B, and eukaryotic translation initiation factor 4E-binding protein 1.
Time Frame: Up to day 15 of course 1
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Days on Therapy
Description: Percentage of days on therapy will be calculated using the formula: (expected - actual days)/expected x 100.
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

5. Secondary Outcome: Dose Interruptions and Adjustments
Description: Dose interruptions and adjustments will be made on a per subject basis and total for the population.
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

6. Secondary Outcome: Frequency of Treatments for Stomatitis
Description: Frequency of treatments for stomatitis will be collection of prescription and non-prescription interventions.
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

7. Secondary Outcome: Type of Treatments for Stomatitis
Description: Type of treatments for stomatitis will be collection of prescription and non-prescription interventions.
Time Frame: Up to 6 months
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

8. Secondary Outcome: Response Rate Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Response rate will be measured at different time points, e.g. 8, 16, and 24 weeks, and will be summarized as percentage of stable disease, complete remission or partial remission along with 95% confidence interval.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Real-time Pharmacokinetic TDM of Everolimus) (N=2)
Elevated glucose (Metabolism and nutrition disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Generalized acne (Skin and subcutaneous tissue disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Trial closed early due to lack of timely accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes